CLINICAL TRIAL: NCT04532866
Title: Brain Changes and Spatial Navigation After Long-Duration Isolation and Confinement and the Significance of Virtual Earth Gazing to Augment Sensory Stimulation
Brief Title: Brain Changes in Response to Long-Duration Isolation and Confinement
Acronym: BRAIVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: The Institute of Biomedical Problems (IBMP) (Unknown); National Aeronautics and Space Administration (NASA) (U.S. Federal Agency); European Space Agency (Other); Max Planck Institute for Human Development (Other); Simon Fraser University (Other); University of California (Other); University of York (Other)
Responsible Party: Principal Investigator, Alexander C. Stahn, Principal Investigator, Charite University, Berlin, Germany
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 400118
Record Dates: First submitted 2020-08-19; First posted 2020-08-31 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Isolation, Social; Virtual Reality; Spatial Navigation
Keywords: Sensory deprivation; Spaceflight; Social isolation; Spatial navigation
MeSH Terms: conditions — Social Isolation; Spatial Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isolation and Confinement (Experimental): Six crew members will spend 8 months isolated and confined in the spaceflight analog NEK in Moscow.
  Interventions: Behavioral: Isolation and Confinement
- Control Group (No Intervention): Up to ten participants matched for age, gender, and educational background undergo the same test protocol as the experimental group at identical points in time but without being isolated and confined in the NEK facility.

INTERVENTIONS:
Behavioral: Isolation and Confinement — Eight months of isolation and confinement in the spaceflight analog NEK in Moscow
  Arms: Isolation and Confinement

SUMMARY:
This study investigates the time course and magnitude of eight months of isolation and confinement in a spaceflight analog facility on brain changes and cognitive performance. The study also assesses the feasibility of an immersive and interactive virtual environment (VE) to enhance positive affect and mental well-being during prolonged isolation and confinement.

DETAILED DESCRIPTION:
The study investigates the neurobehavioural risks associated with future exploratory space missions and their mitigation as part of the isolation and confinement program "SIRIUS" (Scientific International Research In Unique terrestrial Station). The overarching objective of the study is two-fold.

The first objective is to investigate the time course and magnitude of eight months of isolation and confinement in the spaceflight analog facility "NEK" at the Institute of Biomedical Problems (IBMP) in Moscow on brain changes, cognitive performance, and biochemical adaptations, and compare these data to a sex- and age-matched control group. To achieve this aim, multi-modal magnetic resonance imaging (MRI) data before and after the intervention to assess structural and functional brain changes before, and after the experiment will be collected. Furthermore, cognitive performance using a series of computer-based tests will be determined and blood and saliva samples to identify biochemical changes associated with brain plasticity and learning before, during, and after the experiment will be collected.

Second, to address the need for sensory stimulation countermeasures during prolonged isolation and confinement, the feasibility of a highly immersive and interactive virtual environment (VE) to enhance positive affect and mental well-being will be assessed. To achieve this aim, the acute physiological and behavioral effects associated with the proposed sensory augmentation measure will be quantified (Does VE elicit immediate physiological and/or behavioral changes during long-duration isolation and confinement?). It will be verified whether there is an adaptation to the experience with repeated exposure bouts (Can VE elicit similar physiological and or behavioral responses after the VE exposure has been administered recurrently?). The administration rate is optimized relative to crew burden/compliance and scientific return (one administration once a month). This will also ensure that the approach will not have any chronic effects interfering with the primary outcomes of the first objective or any countermeasures foreseen by IBMP. These data will provide essential insights about the efficacy of a new, highly immersive, and target specific VR-based sensory stimulation augmentation to mitigate some of the risks associated with sensory monotony and visual disconnection from Earth during exploration-type missions. The two objectives will deliver a highly unique and comprehensive set of integrated neuroimaging and neurocognitive tools for the evaluation and ultimately prevention of adverse effects on brain plasticity and behavior.

ELIGIBILITY:
Inclusion Criteria:

* Candidates who are professionals in the aerospace industry or related fields are eligible at a lower age limit of 28
* Height not to exceed 180 cm.
* Willing to be confined and isolated for up to 8 months.
* English and Russian verbal and written proficiency not lower than intermediate
* Absence of chronic disease or psychological deviations

Exclusion Criteria:

* Everybody who does not meet listed above requirements
* Past mental, cardiovascular, musculoskeletal and/or neurovestibular disorders or diseases
* Pronounced orthostatic intolerance or vestibular balance disorders (kinetosis)
* Abuses of drugs, medication or alcohol
* Claustrophobia
* Malnutrition up to 6 months before the start of the study
* Intake of anabolic steroids up to 6 months before study initiation
* Metal implants or other osteosynthesis materials
* Bisphosphonate therapy
* Taking medication that could influence the results of the examination.
* Taking hormonal contraceptives in the last 6 months before the start of the study
* Menstrual disorders
* Delivery up to 6 months before the start of studies
* clinically manifest abnormalities in the resting ECG that preclude participation in the study
* Hypertension (> 130/85 mmHg)
* Increased risk of thrombosis
* Increased risk of stroke
* Infection with HIV or HBV
* HIV, hepatitis A, B, or tuberculosis infection
* clinically manifest changes in the differential blood count
* Clinically manifest changes according to the Comprehensive Metabolic Panel (CMP) (blood urea, uric acid, creatinine, total bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), Alkaline Phosphatase (ALP), L-Lactate dehydrogenase (LDH), Glutamyltransferase (GGT), sodium, potassium, chloride, phosphorus, calcium, magnesium, CO2, total protein, albumin, globulin, fasting glucose (< 100mg/dL)
* clinically manifest iron deficiency: < 10 mg/L or < 20 mg/L for women and men respectively
* clinically manifest lipid metabolism disorders
* clinically manifest vitamin D deficiency
* clinical manifest increase of C-reactive protein
* Tuberculosis infection
* Gastroesophageal reflux
* Ulcers
* Kidney disease and/or kidney stones
* Thyroid dysfunction
* Tinnitus
* Sensorineural hearing loss from 30 dB
* Pacemaker or internal defibrillator
* metallic implants (e.g. orthopaedic plates after bone fractures, joint replacement, surgical clips or staples, artificial heart valves, vein filters)
* metallic splinters (e.g. after an accident or because of war injury)
* non-removable braces
* Tattoos with unknown color composition
* Permanent Make-up
* Cochlear implant (implanted hearing aid)
* Medication pump
* Acupuncture needles
* Any other condition which, in the opinion of the investigator, renders the subject unfit for inclusion in the study

Ages: 28 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in brain structure | pre-intervention, immediately after the intervention, up to 30 days after study completion
  Change in gray matter (whole brain and hippocampus) using magnetic resonance imaging (MRI).
Change in brain function | pre-intervention, immediately after the intervention, up to 30 days after study completion
  Change in BOLD signal using functional magnetic resonance imaging (fMRI).
Change in cognitive performance | pre-intervention, monthly during the intervention, immediately after the intervention, up to 30 days after study completion
  Change in reaction time, accuracy, spatial updating, path integration, visuo-spatial memory and learning, spatial orientation ability, and navigation strategy preferences using a cognitive test battery.
Change in biochemical parameters | pre-intervention, monthly during the intervention, immediately after the intervention, up to 30 days after study completion
  Percent change in BDNF, IGF-1, VEGF, oxytocin, and neurofilament light chain using serum, plasma and EDTA samples.
Change in stress response | pre-intervention, monthly during the intervention, immediately after the intervention, up to 30 days after study completion
  Percent change in salivary cortisol using a cotton swab system.

SECONDARY OUTCOMES:
Biochemical parameters in response to sensory stimulation | Baseline, monthly during the VR intervention, immediately after each VR intervention, and up to 1h after the VR intervention
  Assessing whether percent of salivary cortisol and the biochemical parameters BDNF, IGF-1, VEGF, oxytocin, and neurofilament light chain change in response to a sensory stimulation using virtual reality (VR).
Markers of mood and mental well-being in response to sensory stimulation | pre-intervention, monthly during VR stimulation, monthly immediately after VR stimulation, monthly up to 1h after VR stimulation
  Assessing by means of Visual Analog Scales whether subjective markers of mood and mental well-being change in response to sensory stimulation using virtual reality (VR).

OTHER OUTCOMES:
Correlation between changes in brain structure and function and changes in cognitive performance | pre-intervention, monthly during the intervention, immediately after the intervention, up to 30 days after study completion
  Correlation between changes in brain structure and function and changes in reaction time, accuracy, spatial updating, path integration, visuo-spatial memory and learning, spatial orientation ability, and navigation strategy preferences.
Correlation between changes in brain structure and function and changes in biochemical parameters | pre-intervention, monthly during the intervention, immediately after the intervention, up to 30 days after study completion
  Correlation between changes in brain structure and function and changes in BDNF, IGF-1, VEGF, oxytocin, and neurofilament light chain.
Correlation between changes in cognitive performance and changes in biochemical parameters | pre-intervention, monthly during the intervention, immediately after the intervention, up to 30 days after study completion
  Correlation between changes in reaction time, accuracy, spatial updating, path integration, visuo-spatial memory and learning, spatial orientation ability, and navigation strategy preferences and changes in BDNF, IGF-1, VEGF, oxytocin, and neurofilament light chain.
Correlation between changes in biochemical parameters and markers of mood and mental well-being in response to sensory stimulation | pre-intervention, monthly during VR stimulation, monthly immediately after VR stimulation, monthly up to 1h after VR stimulation
  Correlation between changes in percent of salivary cortisol and BDNF, IGF-1, VEGF, oxytocin, and neurofilament light chain and markers of mood and mental well-being assessed by Visual Analog Scales in response to sensory stimulation using virtual reality (VR).

CONTACTS AND LOCATIONS:
Overall Officials: Alexander C Stahn, PhD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- NEK, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No